CLINICAL TRIAL: NCT03037216
Title: Investigation of Exercise Training-Induced Myokines and Adipolkines in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-34
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Healthy
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Exercise-Training Intervention (Experimental): Subjects will undergo a 10-week aerobic exercise protocol.
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — 10 Week aerobic exercise training

SUMMARY:
The purpose of this study is to find out whether exercise training leads to changes in the blood that are produced by exercised muscles and if these changes produce new hormones that affect the body's regulation of sugar and body weight.

ELIGIBILITY:
Inclusion Criteria:

- Age between 18-35. Body mass index (BMI) must be ≥18.5 and ≤27 kg/m2. HbA1c values ≤5.7%

Exclusion Criteria:

* Age <18 and >50
* HbA1c ≥ 5.7%; heart or lung disease
* acute systemic infection accompanied by fever, body aches, or swollen lymph glands
* BMI > 27 kg/m2
* current dieting or weight loss efforts
* current pregnancy or breastfeeding
* known history of HIV/AIDS; cancer
* biochemical evidence of renal or hepatic dysfunction; renal or liver disease demyelinating diseases such as multiple sclerosis or amyotrophic lateral sclerosis
* recent blood donation
* clinical history of stroke
* hypertension (systolic > 140 mmHg or diastolic > 90 mmHg)
* type 1 or 2 diabetes; inability to exercise at 50% of predicted heart rate (HR) reserve at baseline
* Participants taking beta-blockers Participants who screen positive for The American Heart Association's contraindications to exercise testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Changes in circulating proteins in the blood. | Baseline vs. Post 10 Week Training.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Goodyear, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No